CLINICAL TRIAL: NCT05799482
Title: pATienT ExperieNces wiTh covId fOllow-up Clinic
Brief Title: Exploring the Experiences, Expectations and Preferences of Patients With the UHS COVID-19 Follow-up Clinic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RHM MED1959
Record Dates: First submitted 2023-04-04; First posted 2023-04-05 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cross-sectional arm: One-to-one semi-structured interviews will be conducted with patients who have received care in the UHS COVID follow-up clinics in no more than 12 months prior to study enrolment. Interviews will be conducted at one time point
  Interventions: Other: Qualitative Interview
- Prospective, longitudinal arm: One-to-one semi-structured interviews will be conducted with patients with confirmed prior COVID-19 infection who are scheduled to receive care in the UHS COVID follow-up clinics. Interviews will be conducted before attending the first clinic appointment (baseline) and after discharge from the clinic (at 12 weeks).
  Interventions: Other: Qualitative Interview

INTERVENTIONS:
Other: Qualitative Interview — Qualitative, semi-structured interview

SUMMARY:
People who are older, those who had underlying other health conditions and people living in poorer communities are at increased risk of complications and worse outcome from COVID-19. They are more likely to be admitted to hospital with this virus. In the UK in 2020, over 130,000 people were admitted to hospital with COVID-19. Whilst admission rates fell since then, there is a need to understand better the potential impact of the many symptoms resulting from a COVID-19 infection on patients and the health services. To achieve this, the respiratory team in the University Hospital set up a COVID-19 follow-up clinic for patients who had COVID-19 infection. In this clinic, for a period of 12 weeks patients have chest X-rays, blood tests and virtual medical consultations. The clinic has been running for three years.

This study will be conducted study to understand the expectations, preferences and experiences of patients who have been receiving care in the clinic. On one hand, patients who have received care in the clinic during the last yearwill be interviewed. On the other hand, patients who have been newly referred to the clinic will be interviewed before they start it and also after 12 weeks about how their expectations have been met. Patients will be identified by their clinical team and after consenting to take part in the study, they will be interviewed by qualitative researchers who will also analyse the interview data using scientific methods. The results of this study will help understanding whether changes are to be made to this clinic and also inform future similar services should they be needed.

DETAILED DESCRIPTION:
The long-term consequences of COVID-19 remain unclear. People who are older, have medical comorbidities and those who live in areas of increased socio-economic deprivation are at increased risk of poor outcome and complications from COVID-19 (1).

In 2020, over 130,000 people have been admitted to hospital with COVID-19 in the UK (2). Whilst admission rates fell, the potential impact of 'post-COVID' syndromes on patients and the health services need longer-term further investigation.

The British Thoracic Society (BTS) COVID-19 Guidance advises follow-up of patients who had COVID-19, depending on whether the patient required intensive/higher care versus ward/community care.1. For mild/moderate disease, BTS recommends virtual follow-up with a chest X-ray (1). A wide range of symptoms and reduced HRQoL has been detected in these patients reinforcing the importance of a implementing a holistic approach advocated by the BTS and other guidelines (2).

The COVID follow-up service was set up in 2020 in the Southampton General Hospital to provide longer-term care to patients with COVID-19 chest symptoms. The changing nature of the pandemic and an extension of the cohort from patients discharged after hospital stay for COVID-19 infection to previously not hospitalised patients referred by GPs call for an evaluation of the COVID follow-up clinic to explore patient experiences, expectations, and preferences with this service.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Must have had a diagnosis of COVID-19 infection
* Must have been discharged from hospital following admission with Covid-19 infection OR
* Must have been referred to by their GP and accepted into the UHS COVID follow-up clinic
* Retrospective study arm: must have been receiving care in the UHS COVID follow-up clinic at any stage in the last 12 months
* Prospective study arm: must be newly referred to UHS COVID follow-up clinic
* Conversational level of English that does not require a translator
* Giving written informed consent

Exclusion Criteria:

* Less than 18 years old
* Not followed up at UHS post discharge from hospital after admission for COVID-19 infection OR
* Not accepted into the UHS COVID follow-up clinic
* Retrospective study arm: received care in the COVID follow-up clinic more than 12 months prior to enrolment in the study
* Unwilling or unable to give informed consent
* Unwilling or unable to participate in the interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The research population of interest for this study is patients followed up in the UHS COVID follow-up clinic following diagnosed COVID-19 infection. This will include all patients deemed appropriate by their clinical team to receive this clinical service
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Qualitative Interview | 12 months
  Experiences, preferences and expectations of patients receiving care in the UHS COVID-19 follow-up clinic

CONTACTS AND LOCATIONS:
Locations (1):
- Judit Varkonyi-Sepp, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Throughout the study, the researchers will be working with the Public and Patient Involvement group to develop a dissemination strategy of the results to the study participants and other stakeholders and/or the public as appropriate.

REFERENCES:
- [Background] George PM, Barratt SL, Condliffe R, Desai SR, Devaraj A, Forrest I, Gibbons MA, Hart N, Jenkins RG, McAuley DF, Patel BV, Thwaite E, Spencer LG. Respiratory follow-up of patients with COVID-19 pneumonia. Thorax. 2020 Nov;75(11):1009-1016. doi: 10.1136/thoraxjnl-2020-215314. Epub 2020 Aug 24. PMID 32839287
- [Background] Arnold DT, Hamilton FW, Milne A, Morley AJ, Viner J, Attwood M, Noel A, Gunning S, Hatrick J, Hamilton S, Elvers KT, Hyams C, Bibby A, Moran E, Adamali HI, Dodd JW, Maskell NA, Barratt SL. Patient outcomes after hospitalisation with COVID-19 and implications for follow-up: results from a prospective UK cohort. Thorax. 2021 Apr;76(4):399-401. doi: 10.1136/thoraxjnl-2020-216086. Epub 2020 Dec 3. PMID 33273026
- [Background] Wallis TJ, Welham B, Kong A, Morelli T, Azim A, Horno J, Wilkinson M, Burke H, Freeman A, Wilkinson TM, Jones MG, Marshall BG. Predicting the risk of chest radiograph abnormality 12-weeks post hospitalisation with SARS CoV-2 PCR confirmed COVID-19. Respir Res. 2022 Oct 31;23(1):297. doi: 10.1186/s12931-022-02217-0. PMID 36316730
- [Background] Wallis TJM, Heiden E, Horno J, Welham B, Burke H, Freeman A, Dexter L, Fazleen A, Kong A, McQuitty C, Watson M, Poole S, Brendish NJ, Clark TW, Wilkinson TMA, Jones MG, Marshall BG. Risk factors for persistent abnormality on chest radiographs at 12-weeks post hospitalisation with PCR confirmed COVID-19. Respir Res. 2021 May 21;22(1):157. doi: 10.1186/s12931-021-01750-8. PMID 34020644
- See also: HRA amendment guidance — http://www.hra.nhs.uk/resources/after-you-apply/amendments/